CLINICAL TRIAL: NCT06329934
Title: Effect of Refined Nursing in Rehabilitation Training for Patients With Brain Injury During the Recovery Period: An Observational Study
Brief Title: Refined Nursing in Rehabilitation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinxiang Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XXZY-003
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2022-05

CONDITIONS: Brain Injuries
Keywords: Refined nursing; Coma; Rehabilitation training
MeSH Terms: conditions — Brain Injuries; Coma | interventions — Methods; Humidity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): Establishment of a hierarchical monitoring and management team, Assessment of pressure injury, Communication, Intervention for pressure ulcer, Rehabilitation training
  Interventions: Behavioral: Establishment of a hierarchical monitoring and management team; Behavioral: Assessment of pressure injury; Behavioral: Communication; Behavioral: Intervention for pressure ulcer; Behavioral: Rehabilitation training
- the control group (Active Comparator): timely introduction of the current patient's condition to family members to alleviate their concerns, maintaining appropriate temperature (20 ℃~22 ℃) and humidity (60.0%~70.0%) in the ward, careful observation of vital signs such as heart rate, blood oxygen saturation, and blood pressure in patients, rehabilitation training
  Interventions: Behavioral: Rehabilitation training; Behavioral: introduction of the current patient's condition to family members; Behavioral: maintaining appropriate temperature and humidity in the ward; Behavioral: careful observation of vital signs in patients

INTERVENTIONS:
Behavioral: Establishment of a hierarchical monitoring and management team — To be specific, the head nurse served as the team leader to conduct comprehensive macro supervision; moreover, there were 3 responsible team leaders and 6 responsible nurses, all of whom had rich clinical nursing experience and solid theoretical knowledge of pressure injury. Consequently, a joint-action mechanism of the head nurse - responsible team leader - responsible nurses was developed to facilitate the unification of the training of nursing content, precautions, etc.
  Arms: the intervention group
Behavioral: Assessment of pressure injury — Based on the postoperative coma of patients, the Braden assessment scale was applied to effectively evaluate patients from six dimensions of sensory perception, moisture, activity mode, mobility, nutrition, friction, and shear. The total score was 23 points. Patients scoring 13~14 points were evaluated by Braden once per week; and those scoring ≤12 points were evaluated at a frequency of 3d/ time.
  Arms: the intervention group
Behavioral: Communication — Through intensive face-to-face communication with family members, timely information on the surgical effect, mechanism of pressure injury, preventive measures, and clinical manifestations through intuitive methods such as PPT and video, family members were taught with basic knowledge of pressure injury, and guided to inform medical staff in a timely manner when patients had symptoms of pressure ulcer. Simultaneously, by case sharing and positive suggestions, family members were supported to alleviate their concerns and improve their coordination with treatment
  Arms: the intervention group
Behavioral: Intervention for pressure ulcer — For patients with a Braden score of >14 points, attention should be paid to keeping skin dry and clean, regularly changing bed sheets and bedding (once per day). Patients with Braden score of 13-14 points should be provided with sponge mattresses, increased times of turning over once per 2 hours, and soft pillows or foam dressings at the site of occipital protuberance to relieve pressure and prevent pressure injury. For patients with Braden score ≤12 points, medical staff should repeatedly emphasize to their families the harm of pressure injury to postoperative recovery.
  Arms: the intervention group
Behavioral: Rehabilitation training — After regaining consciousness with stable vital signs, patients received rehabilitation training following the principle of association of activity and inertia in a regular order. Patients were guided to perform upper limb movements, joint flexion, lower limb flexion and extension, as well as daily training such as washing face, rinsing mouth, and dressing at a frequency of 3~4 times/d. Moreover, patients were advised to minimize violent behaviors such as laughing and talking loudly
Behavioral: introduction of the current patient's condition to family members — timely introduction of the current patient's condition to family members to alleviate their concerns
  Arms: the control group
Behavioral: maintaining appropriate temperature and humidity in the ward — maintaining appropriate temperature (20 ℃~22 ℃) and humidity (60.0%~70.0%) in the ward
  Arms: the control group
Behavioral: careful observation of vital signs in patients — careful observation of vital signs such as heart rate, blood oxygen saturation, and blood pressure in patients
  Arms: the control group

SUMMARY:
This study is to explore the clinical effect of refined nursing in rehabilitation training for patients with brain injury during the recovery period. Patients in the control group were provided with routine nursing intervention, while patients in the study group adopted a nursing mode based on the concept of refinement treatment. Comparison was made in terms of the Glasgow Coma Scale (GCS) score, cognitive function score, functional independence score, nursing satisfaction, and incidence of complications.

DETAILED DESCRIPTION:
This study is to explore the clinical effect of refined nursing in rehabilitation training for patients with brain injury during the recovery period. The subjects of the study were 96 patients with severe traumatic brain injury (TBI). According to the order of visits, there were 48 patients in the study group and the control group, respectively.Patients in the control group were provided with routine nursing intervention, while patients in the study group adopted a nursing mode based on the concept of refinement treatment. Comparison was made in terms of the Glasgow Coma Scale (GCS) score, cognitive function score, functional independence score, nursing satisfaction, and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with severe TBI through imaging examinations such as head CT and magnetic resonance imaging
* patients with surgical indications
* patients with Glasgow Coma Scale (GCS) ≤8 points
* patients with complete clinical data
* patients with written informed consent provided by family members

Exclusion Criteria:

* patients with organic lesions of major organs such as liver and kidney
* patients with contraindications for surgery
* patients with primary diseases such as cerebral hemorrhage and cerebral infarction
* patients with combined or multiple injuries
* patients with respiratory failure
* patients whose family members had cognitive impairment or abnormal mental behaviors

Ages: 33 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
GCS scores | one day before the intervention
  The highest GCS score was 15 points, indicating clear consciousness; while patients with 13-15, 9-12, and ≤8 points were classified as mild, moderate consciousness disorder, and coma, respectively. Patients with lower scores might indicate more serious consciousness disorder
GCS scores | 2 months after rehabilitation treatment
  The highest GCS score was 15 points, indicating clear consciousness; while patients with 13-15, 9-12, and ≤8 points were classified as mild, moderate consciousness disorder, and coma, respectively. Patients with lower scores might indicate more serious consciousness disorder
cognitive function scores | one day before the intervention
  Cognitive function was evaluated using the Chinese version of the Neurobehavioral Cognitive Status Exam (NCSE) to assess the cognitive function of patients before and 2 months after rehabilitation treatment. This scale includes 10 items, i.e., spatial orientation (12 points), concentration (8 points), understandability (6 points), retelling (12 points), naming (8 points), spatial construction (6 points), memory (12 points), computing (4 points), similarity (8 points), and judgment (6 points)
cognitive function scores | 2 months after rehabilitation treatment
  Cognitive function was evaluated using the Chinese version of the Neurobehavioral Cognitive Status Exam (NCSE) to assess the cognitive function of patients before and 2 months after rehabilitation treatment. This scale includes 10 items, i.e., spatial orientation (12 points), concentration (8 points), understandability (6 points), retelling (12 points), naming (8 points), spatial construction (6 points), memory (12 points), computing (4 points), similarity (8 points), and judgment (6 points)
functional independence scores | one day before the intervention
  Functional Independence Measure (FIM), utilizing a 7-point ordinal scale, was employed to assess the functional independence of two groups of patients before and 2 months after rehabilitation treatment. FIM measures independent performance in self-care, sphincter control, mobility, locomotion, communication, social cognition, etc. The minimum score is 18 points, and the maximum score is 126 points (91 points for motor function and 35 points for cognitive function)
functional independence scores | 2 months after rehabilitation treatment
  Functional Independence Measure (FIM), utilizing a 7-point ordinal scale, was employed to assess the functional independence of two groups of patients before and 2 months after rehabilitation treatment. FIM measures independent performance in self-care, sphincter control, mobility, locomotion, communication, social cognition, etc. The minimum score is 18 points, and the maximum score is 126 points (91 points for motor function and 35 points for cognitive function)
Newcastle Satisfaction with Nursing Scale (NSNS) | one day before the intervention
  The Newcastle Satisfaction with Nursing Scale (NSNS) was used to survey patient's nursing satisfaction. This scale measures patient's satisfaction with nursing care from 19 items, including nurse work ability, communication attitude, psychological counseling, nursing support, safety management, etc. It uses a 1-5 point scoring system, with a maximum possible score of 19-95 points. A score of ≥77, 58~76, 39~57 and ≤38 points indicated very satisfied, satisfied, somewhat satisfied, and dissatisfied, respectively. Satisfaction rate= (Cases of very satisfied + satisfied + somewhat satisfied)÷total cases
Newcastle Satisfaction with Nursing Scale (NSNS) | 2 months after rehabilitation treatment
  The Newcastle Satisfaction with Nursing Scale (NSNS) was used to survey patient's nursing satisfaction. This scale measures patient's satisfaction with nursing care from 19 items, including nurse work ability, communication attitude, psychological counseling, nursing support, safety management, etc. It uses a 1-5 point scoring system, with a maximum possible score of 19-95 points. A score of ≥77, 58~76, 39~57 and ≤38 points indicated very satisfied, satisfied, somewhat satisfied, and dissatisfied, respectively. Satisfaction rate= (Cases of very satisfied + satisfied + somewhat satisfied)÷total cases
incidence of adverse reactions | one day before the intervention
  Incidence (%)=Number of patients with complications/48×100%
incidence of adverse reactions | 2 months after rehabilitation treatment
  Incidence (%)=Number of patients with complications/48×100%

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, Principal Investigator — Xinxiang Central Hospital
Locations (1):
- Effect of Refined Nursing in Rehabilitation Training for Patients with Brain Injury During the Recovery Period: An Observational Study, Xinxiang, Henan, China